CLINICAL TRIAL: NCT04803123
Title: Window Trial to Evaluate Molecular Response to PI3K Inhibition With Copanlisib in Relapsed or Refractory Adult B-cell Acute Lymphoblastic Leukemia
Brief Title: Window Trial to Evaluate Molecular Response to PI3K Inhibition With Copanlisib in r/r Adult B-cell ALL
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Sponsor halted clinical development of study drug
Sponsor: Dorothy Sipkins, MD, PhD (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor-Investigator, Dorothy Sipkins, MD, PhD, Associate Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00105967
Record Dates: First submitted 2021-03-15; First posted 2021-03-17 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Leukemia, Acute Lymphocytic
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — copanlisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Copanilisib (Experimental)
  Interventions: Drug: Copanlisib

INTERVENTIONS:
Drug: Copanlisib — Patients must receive at least one dose of copanlisib prior to standard therapy to be evaluable.

SUMMARY:
This study will provide an evaluation of biologic markers of leukemia cell response following a single dose of copanlisib prior to any salvage induction therapy in a projected cohort of 10 relapsed/refractory B-ALL patients.

ELIGIBILITY:
Inclusion Criteria:

1. Relapsed/refractory, Philadelphia chromosome positive or negative, B-cell, adult (≥ age 18) acute lymphoblastic leukemia (including bone marrow, extramedullary, CNS disease, or all), with or without prior hematopoietic stem cell transplant.

   Philadelphia chromosome positive patients prior to enrollment must have documented treatment failure to all FDA-approved for use in R/R ALL tyrosine kinase inhibitor (TKI) therapy, or have previously been deemed by their treating physician to not be a candidate for further TKI therapy.
2. ECOG 0-3.
3. CrCl ≥ 30 mL/minute.
4. Bilirubin ≤ 1.5x upper limit of normal (ULN), AST/ALT ≤ 3x ULN.
5. Any patients with known pulmonary disease (including COPD, asthma, ongoing tobacco use, pulmonary hypertension, pulmonary sarcoidosis, or other relevant pulmonary disease which severely limits their pulmonary function), require an assessment of lung capacity with pulmonary function testing prior to acceptance to the study, with a threshold acceptance of DLCO > 40% corrected.

Exclusion Criteria:

1. History of or concurrent condition of interstitial lung disease or autoimmune pneumonitis.
2. Active pneumonia requiring treatment, including Pneumocystis jirovecci pneumonia (PJP).
3. History of type 1 diabetes mellitus.
4. Type 2 diabetes mellitus with HgbA1C ≥10% while on treatment for diabetes.
5. Uncontrolled hypertension despite optimal medical management (per investigator's assessment).
6. Untreated human immunodeficiency virus (HIV).
7. Active replication of hepatitis B or active hepatitis C. Those with prior disease who are PCR negative at enrollment and meet liver function eligibility criterion are eligible.
8. Cytomegalovirus (CMV) infection with positive PCR at baseline. CMV PCR test is considered positive if the result can be interpreted as a CMV viremia according to institutional standard.
9. History of hematopoietic stem cell transplant with active GVHD requiring > 10 mg of prednisone daily or equivalent.
10. History of calcineurin inhibitor use in the last 28 days prior to enrollment.
11. Patients requiring immediate cytoreductive therapy. Exceptions for: patients whose peripheral blast counts are being controlled by single agent or combination therapy with steroids and/or hydroxyurea.
12. Pregnancy.
13. Active concurrent malignancy requiring ongoing treatment. Exceptions for: resected breast cancer being treated with hormonal therapy only, prostate cancer treated with hormonal therapy not progressing within the past year, if subject has received definitive local therapy (i.e., surgical excision, external beam radiation, or other local therapy with curative intent), non-melanoma skin cancers, or carcinoma in situ.
14. Active COVID-19 infection.
15. Progressive and/or uncontrolled infections despite active treatment.
16. Patients with residual toxicities related to prior treatment (including chemotherapy, immunotherapy, clinical trial, surgery, radiotherapy, or hematopoietic stem cell transplant) persistently > Grade 1 despite adequate treatment. Exceptions for: patients with residual toxicity related to prior treatment of ≤Grade 2 which is stable prior to enrollment and for which the natural history would not be expected to change over time; toxicity which cannot be reasonably excluded to be due to disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2023-04-03 (Actual); Study Completion 2023-04-26 (Actual)

PRIMARY OUTCOMES:
Evaluate the effect of copanlisib exposure on alpha-6 integrin expression levels in leukemic blasts using flow cytometry. | 1 year

SECONDARY OUTCOMES:
Evaluate the effect of copanlisib exposure on proliferation of ALL blasts as determined by flow cytometric blast cell Ki-67 index. | 1 year
Evaluate the effect of copanlisib exposure on proliferation of ALL blasts as determined by peripheral blood hematologic parameters (CBC and WBC differential including blast percentage). | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy Sipkins, MD, Principal Investigator — Duke University
Locations (1):
- Duke Cancer Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No